## The Effect of Gastric Acid Suppression on Probiotic Colonization

## Statistical Analysis Plan NCT03327051

December 13, 2019

The relative percentage abundance was obtained by summing the levels of VSL#3 probiotic strains detected in the study samples. Statistical analysis was performed using GraphPad prizm. Two-way ANOVA with Bonferroni posttest was used for multi-variable analyses (within-group differences between week 0 and week 4). A p-value of <0.05 would be considered statistically significant.